CLINICAL TRIAL: NCT02123303
Title: The Incidence of Orthostatic Hypotension Among Veterans
Brief Title: Orthostatic Hypotension Among Veterans
Acronym: OH
Status: Completed | Type: Observational
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jill M. Wecht, Ed.D., Research Health Science Specialist, James J. Peters Veterans Affairs Medical Center
Other Study IDs: WEC-10-038
Record Dates: First submitted 2014-04-23; First posted 2014-04-25 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Hypotension, Orthostatic Hypotension
Keywords: Hypotension, Orthostatic Hypotension
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Veterans

SUMMARY:
Orthostatic hypotension (OH) is defined as a fall in blood pressure when standing. Several different underlying diseases, conditions, or combinations of medicines may contribute to OH; therefore the cause of the condition varies among individuals. Some studies have shown that OH is associated with an increase in the rate of death, but it is not clear what role OH plays in increased morbidity. By studying what the prevalence of OH is in a generalized veteran population we expect increase clinical awareness of the degree of the problem so that patient care might be improved.

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* Between the ages of 18 and 89

Exclusion Criteria:

* Current illness/infection
* Pregnant

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any able-bodied veteran (able to independently stand for 10 minutes) that presents for a routine clinical visit or a neurological clinic visit at the James J. Peters VA Medical Center and does not have an acute illness or infection is eligible to participate in the study.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure from supine to standing. | Eval#1: 10min supine; Eval#2: 10min standing;
  Change in blood pressure between Evaluation #1 and Evaluation #2.

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Wecht, EdD, Principal Investigator — James J. Peters VAMC
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States